CLINICAL TRIAL: NCT02295241
Title: Improving Muscle Assessment in Older Adults - The "Can We Build a Better Mouse Trap?" Study
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-1109
Record Dates: First submitted 2014-10-03; First posted 2014-11-20 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Sarcopenia
Keywords: Sarcopenia, muscles, aging
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be drawn to obtain a serum chemistry panel to document health status of the study participants. For subjects who agree to optional banking, serum aliquots will be obtained and banked for future study of markers relevant to musculoskeletal health.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — This is an observational trial, no interventions are being used.

SUMMARY:
The primary aim of this study is to compare traditional muscle function tests with computerized versions using body-worn motion sensors and video motion analysis of the same tests. The investigators selected the Timed Up and Go (TUG) test as the investigators primary variable for this aim with several other function tests (e.g., repeated chair rise, 6-meter walk, 2-minute walk, Romberg stance, semi-tandem / tandem stance) as secondary variables. The investigators primary hypothesis is that the computerized versions of the TUG test are highly correlated (>0.9) with the traditional method, but with comparable or better reproducibility. Secondary analyses will correlate other function tests with their computerized version, again with the hypothesis that they are highly correlated and that computerized versions are of similar or better reproducibility. This analysis will also compare traditional assessments of balance with a computerized balance method, computerized dynamic posturography.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory, community dwelling men and women age ≥ 70 years
2. Able and willing to sign informed consent
3. Able to stand without assistance

Exclusion Criteria:

1. History of myocardial infarction within the prior six months or ongoing angina
2. History of injury or surgery within the prior six months which limits the ability to ambulate
3. History of malignancy with metastasis to the musculoskeletal system
4. Neuromuscular disease or severe end organ disease impairing balance or muscle function to the degree that completion of all study tests is unlikely.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will evaluate community dwelling women and men ≥ 70 years recruited from the Madison, Wisconsin area.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The comparison of results of traditional physical function tests with the results of computerized versions (body worn sensors and Kinect system) of the same tests. | All physical function tests will be performed at the first visit and visit 2 up to 4 days later
  Short-term reproducibility of traditional vs. computerized functional tests will also be compared.

SECONDARY OUTCOMES:
Explore the capabilities of the Microsoft Kinect system to record and analyze muscle function tests and correlate the Microsoft Kinect system to a gold standard motion analysis system. | All physical function tests will be performed at the first visit and visit 2 up to 4 days later.
Validate the use of BIS (Bioelectrical Impedance Spectroscopy) to adjust DXA (Dual Energy X-ray Absorptiometry) -measured body composition by providing muscle mass measurement | BIS is performed at visit 1 and visit 2 up to 4 days later. DXA is performed at visit 2.
  The relationship of lean mass, as estimated by DXA and BIS with muscle mass as measured by deuterated creatine dilution as a nominal gold standard. Additionally, the correlation of lean mass as measured by DXA and muscle mass as measured by BIS and creatine dilution with muscle function tests.
Correlate various ratios of lean or muscle mass / DXA measured fat mass with functional tests. | All physical function tests will be performed at the screen and follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Binkley, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison Osteoporosis Clinical Research Program, Madison, Wisconsin, United States